CLINICAL TRIAL: NCT03611413
Title: Feasibility and Effects of an Enhanced Recovery vs Conventional Care After Emergency Colon Surgery for Patients With Left Colon Perforation.
Status: Completed | Type: Observational
Sponsor: Antonio Arroyo Sebastian (Other)
Responsible Party: Sponsor-Investigator, Antonio Arroyo Sebastian, DOCTOR, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Other Study IDs: GERM-01-18
Record Dates: First submitted 2018-07-18; First posted 2018-08-02 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Colon Perforation
Keywords: COLON PERFORATION SURGERY

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS programme: Patients who have been treated under an ERAS programm
  Interventions: Procedure: ERAS care
- conventional care: Patients who have been treated under an conventional care

INTERVENTIONS:
Procedure: ERAS care — ERAS PROTOCOL
  Groups: ERAS programme

SUMMARY:
A study was designed with a prospective cohort of all patients undergoing urgent surgery for left colon perforation between March 2014 and June 2017 who were treated according to a specific ERAS programme (ERAS group/29 patients). This group was compared with a historic case-matched control group with conventional care (CC group/21 patients). The main endpoints were postoperative 30-day morbidity, length of postoperative hospital stay, rate of readmission within 30 days, and mortality. The inclusion criteria were patients over 18 years old with a low-moderate risk of mortality according to a Peritonitis Severity Score (PSS) between 6-11 points.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients over 18 years old with a low-moderate risk of mortality according to a Peritonitis Severity Score (PSS), between 6-11 points.

Exclusion Criteria:

* The exclusion criteria were patients under 18 years old and patients with a high risk of mortality according to a PSS equal to or greater than 12 points.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: emergency surgery with a diagnosis of left colon perforation
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
number of items completed of ERAS protocol | 1-month
  to analyze the applicability of a specific ERAS protocol in the management of patients with left colon perforation requiring emergency colon surgery, it will be analyzed the number of items completed of ERAS protocol (YES/NO)